CLINICAL TRIAL: NCT00056719
Title: Genetic Determinants of Ankylosing Spondylitis Severity - Longitudinal Study
Status: Completed | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030131; 03-AR-0131
Record Dates: First submitted 2003-03-21; First posted 2003-03-20 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-12-04

CONDITIONS: Ankylosing Spondylitis
Keywords: Arthritis; Spondylarthropathy; Spine; Hereditary; Disability; Natural History; Ankylosing Spondylitis; Spondyloarthropathy; Spondyloarthritis; AS
MeSH Terms: conditions — Spondylitis, Ankylosing; Arthritis; Spondylarthropathies; Spondylarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will explore how genes may influence the severity of ankylosing spondylitis, a form of arthritis that affects the spine. Patients have inflammation of the joints of the spine, which may cause the bones of the spine to fuse, resulting in difficulty performing daily activities.

Patients who developed ankylosing spondylitis after age 16 may be eligible for this study. The onset of disease is dated to the first appearance of symptoms of inflammatory low back pain or restricted spinal motion. Patients with a spondyloarthropathy other than AS may not participate. Candidates will be screened with a medical history and physical examination, blood test, and review of their medical records. They will also complete a questionnaire about their disease symptoms and medical history.

Those enrolled in the study will return to the NIH Clinical Center at 6, 12, 18, 24, 30, 36, 42, 48, 54, and 60 months after screening for examination of the joints, measurement of flexibility of the spine, and a blood test. They will also complete symptoms assessment and coping questionnaires. At the first study visit (screening visit), x-rays will be taken of the pelvis, lower back, and neck, if recent X-rays (within 1 year) are not available. These x-ray studies will be repeated on all patients every two years during the study (at 24 and 48 months after screening).

DETAILED DESCRIPTION:
The susceptibility to ankylosing spondylitis (AS) is largely genetically determined. Recent studies suggest that the severity of AS is also influenced by genetic factors. The goal of this study is to identify genes that influence the severity of AS. We hypothesize that genetic markers of susceptibility, including human leukocyte antigen (HLA) polymorphisms, and genes that regulate inflammation and bone formation, influence the severity of AS.

In this prospective longitudinal study, we will test the association of several genetic markers with the severity of AS. Approximately 700 patients will be included. Measures of AS severity will be patient-reported pain and stiffness, functional disability, patient and physician global assessments, joint counts, number of tender entheses, spinal mobility, and laboratory measures of inflammation. These measures will be assessed every 6 months for 5 years. We will also evaluate new laboratory tests as measures of the activity of AS.

Identifying genetic markers that are associated with differences in the severity of active inflammation in AS will enhance our understanding of the pathogenesis of this disease by suggesting mechanisms and pathways involved in the development of long-term damage.

ELIGIBILITY:
* INCLUSION AND EXCLUSION CRITERIA:

Participants will:

1. have been diagnosed with AS by the modified New York criteria.
2. be able to read English or Spanish

Potential participants will be excluded if:

1. have a spondyloarthropathy other than AS
2. are unable to provide informed consent
3. anticipate not being available or able to comply with the schedule of study visits

Study entry is not limited by sex or ethnic origin. Children will necessarily be excluded because spondyloarthropathy developing before age 16 is considered a form of juvenile idiopathic arthritis, and because different age-appropriate measures of functional disability and pain would be needed.

Participants will be recruited by physician referral and self-referral. Information about the study will be mailed to local rheumatologists and posted on the NIH website. Notices will also be sent to local chapters of the Arthritis Foundation and the Spondylitis Association of America.

The accrual ceiling will be unlimited. Approximately 700 patients will be enrolled from all study sites. Approximately 150 patients will be recruited at the NIH. Other sites participating in this study are Cedars-Sinai Medical Center, Los Angeles, CA; the University of California-San Francisco, and University of Texas-Houston Health Sciences Center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: identify genes assoc. w/ severity of AS@@@
Sampling Method: Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2003-06-19 (Actual)

PRIMARY OUTCOMES:
identify genes assoc. w/ severity of AS | 10 years
  identify genes assoc. w/ severity of AS

SECONDARY OUTCOMES:
identify genetic polymorphisms of AS
Changes in symptoms of AS over time
Genetic var. in 1st degree rel. of AS pt

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Colbert, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
not yet known

REFERENCES:
- [Background] Boyer GS, Templin DW, Bowler A, Lawrence RC, Everett DF, Heyse SP, Cornoni-Huntley J, Goring WP. A comparison of patients with spondyloarthropathy seen in specialty clinics with those identified in a communitywide epidemiologic study. Has the classic case misled us? Arch Intern Med. 1997 Oct 13;157(18):2111-7. PMID 9382668
- [Background] Mau W, Zeidler H, Mau R, Majewski A, Freyschmidt J, Stangel W, Deicher H. Clinical features and prognosis of patients with possible ankylosing spondylitis. Results of a 10-year followup. J Rheumatol. 1988 Jul;15(7):1109-14. PMID 3262757
- [Background] Amor B, Santos RS, Nahal R, Listrat V, Dougados M. Predictive factors for the longterm outcome of spondyloarthropathies. J Rheumatol. 1994 Oct;21(10):1883-7. PMID 7837155
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2003-AR-0131.html